CLINICAL TRIAL: NCT03906357
Title: Expanded Access of Pemigatinib to Treat a Single Patient With Metastatic Pancreatic Cancer
Status: No longer available | Type: Expanded Access
Sponsor: Incyte Corporation (Industry)
Collaborators: H. Lee Moffitt Cancer Center and Research Institute (Other)
Responsible Party: Sponsor
Other Study IDs: I-54828-20-08
Record Dates: First submitted 2019-04-04; First posted 2019-04-08 (Actual); Last update posted 2022-04-19 (Actual); Status verified 2022-04

MeSH Terms: interventions — pemigatinib

STUDY DESIGN:
Expanded Access Types: Individual

INTERVENTIONS:
Drug: Pemigatinib
  Other Names: INCB054828

SUMMARY:
Expanded access of Pemigatinib to treat a single patient with metastatic pancreatic cancer.

ELIGIBILITY:
Inclusion Criteria:

-

Exclusion Criteria:

-

Age Groups: Child, Adult, Older Adult

CONTACTS AND LOCATIONS:
Overall Officials: Dae Won Kim, MD, Principal Investigator — H. Lee Moffitt Cancer Center and Research Institute